CLINICAL TRIAL: NCT06912360
Title: Use of (Continous Positive Airway Pressure) CPAP in the Management of Acute Hypoxemic Respiratory Failure
Brief Title: Continous Positive Airway Pressure (CPAP) Support for Acute Hypoxemic Respiratory Failure in Burkina Faso
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université NAZI BONI (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Ismael Guibla, Clinical doctor, Université NAZI BONI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSSA 4
Record Dates: First submitted 2025-03-23; First posted 2025-04-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Failure
Keywords: CPAP; Acute hypoxemic respiratory failure; Africa
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: We will have two groups : an interventional group and a standard of care group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP group (Experimental): Continuous CPAP (with Boussignac valve) for the first 6-12 hours, then alternating with standard oxygen therapy. CPAP pressure= 7.5 cmH2O (25L/min) then variations of +/- 2.5 cmH20 according to clinical response and tolerance until weaning from oxygen or presence of intubation criteria
  Interventions: Other: CPAP
- Standard group (No Intervention): Oxygen therapy as required using, simple face masks or high concentration face masks until there are criteria for intubation, or withdrawal from oxygen.

INTERVENTIONS:
Other: CPAP — Continuous Positive Airway Pressure (CPAP) with Boussignac valve
  Arms: CPAP group

SUMMARY:
Acute respiratory failure (ARF) is a frequent medical emergency, involving high costs for health organizations and patients who often require intensive care and respiratory assistance. According to an international study, 61% of hypoxemic patients in intensive care receive invasive ventilation [3]. Invasive mechanical ventilation is often unavailable in low-income countries and non-invasive ventilatory supports such as continuous positive airway pressure (CPAP) and high-flow oxygen therapy (HFO) were very useful during the COVID-19 pandemic. They reduced the rate of intubation and ICU admissions. In addition, CPAP can be used without a ventilator, no electricity is required. So, it could be a support of choice in low-income countries.

Used of Boussignac-type CPAP could potentially reduce the recourse to intubation in patients with acute hypoxemic respiratory failure in a context where access to invasive ventilation remains very limited.

DETAILED DESCRIPTION:
1. Hypothesis :

   The use of Boussignac-type CPAP could reduce the need for intubation in patients with acute respiratory failure in a setting where access to invasive ventilation remains very limited.
2. Objectives

   2.1 Primary Objective

   The primary objective is to evaluate the effect of CPAP use on the occurrence of intubation criteria at 7 days in patients presenting with ARF in the emergency department.

   2.2 Secondary Objectives

   The secondary objectives are:
   * To assess the impact of CPAP use on 28-day mortality in patients with ARF
   * To assess the effectiveness of CPAP use on oxygenation in patients with ARF using the SpO2/FiO2 ratio
   * To assess the impact of CPAP use on hospital stay
   * To assess the safety of CPAP in patients with ARF

   2.3 Ancillary Studies

   The ancillary studies are:
   * To assess the contribution of ultrasound in the management of ARF
   * To determine the etiologies and prognosis of ARF
   * To determine the etiologies and prognosis of patients with ARDS in intensive care
   * To assess the cost of ARF management
3. Methodology 3.1 Study Setting

The Study will take place in the four adult university hospitals in Burkina Faso. Patient recruitment will take place during the same period in the emergency and intensive care departments. Patient inclusion in each hospital will be under the responsibility of an emergency department physician or an anesthesiologist-intensive care physician.

3.2 Study Type

This will be an open-label, multicenter, national randomized clinical trial. The type of oxygenation device does not allow for a blinded study.

3.3 Study Designs

Within 3 hours of validating the inclusion criteria, patients will be assigned to one of the two groups after signing the consent form.

* In both groups, the oxygen flow will be adjusted to achieve an SpO2 of 92% or higher. SpO2 will be measured either using a monitor with integrated SpO2 measurement or using a portable device such as the Lifebox. The remainder of the patient's care will be administered according to the etiology of the ARF at the physician's discretion and according to recommandations. Any omission from the administration of study treatment will be noted on the collection sheet.
* In the standard group Patients assigned to the standard treatment group will receive oxygen delivered via nasal prongs, simple face masks, or a high-concentration face mask (as needed) until intubation criteria are met, death occurs, or oxygen discontinuation criteria are met (an SpO2 greater than 92% without oxygen and a respiratory rate less than 25 breaths/min).

Patients who meet the intubation criteria will either be intubated if a bed and a ventilator are available in intensive care, or may receive, at the discretion of the physician, CPAP treatment as backup treatment in crossover, if invasive ventilation is not possible.

- In the CPAP group Patients assigned to the CPAP plus oxygen group will receive periods of CPAP in addition to standard oxygen therapy. All study centers will use a Boussignac device connected to an oronasal mask consisting of a transparent mask and a soft inflatable cushion. The CPAP pressure level will be determined by the oxygen flow rate according to the correlation table. CPAP will start at 7.5 cmH2O (i.e., a Boussignac supply of 25 L/min). The pressure level will be decreased to 5 cmH2O (i.e., a Boussignac supply of 20 L/min) or increased to 10 cmH2O (i.e., a Boussignac supply of 30 L/min) depending on clinical response and tolerance. For at least the first 6 to 12 hours, CPAP will be administered continuously, then intermittently (for at least 6 hours/day) depending on patient tolerance. CPAP will be continued until endotracheal intubation criteria are met, death occurs, or treatment is discontinued according to the following criteria: SpO2 greater than 92% and respiratory rate less than 25 breaths/min with 3 L of oxygen or less between CPAP sessions. The criteria for discontinuing oxygen administration will be the same as in the standard group.

Patients who meet the intubation criteria will either be intubated if a bed and ventilator are available in intensive care, or will continue CPAP treatment if invasive ventilation is not possible.

3.4 Stratification

Randomization will be stratified by study center and baseline hypoxemia status. Stratification block randomization will be performed using a centralized, secure electronic system.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 years and older will be included in the study if they meet at least one of the following criteria :

* Acute respiratory distress, defined as dyspnea respiratory rate ≥ 25 cycles/min
* Hypoxemia, defined as the need for more 6 liters of oxygen to maintain an oxygen saturation (SpO2) of ≥ 92%. The fraction of inspired oxygen (FiO2) will be estimated using the 3% rule.

Exclusion Criteria:

Patients with any of the following criteria will not be included in the study:

* Pregnant or breastfeeding women
* Persons deprived of their liberty
* Exacerbation of asthma, chronic obstructive pulmonary disease, or another chronic respiratory disease
* Moderate to large amount of unilateral or bilateral undrained pleural effusion
* Contraindication to CPAP: patient refusal, undrained pneumothorax, chest injury, repeated or large vomiting, upper gastrointestinal bleeding, craniofacial trauma, severe upper airway obstruction, or tetraplegia in the initial phase
* Cardiac arrest, severe arrhythmias, shock requiring the use of vasopressors (norepinephrine, adrenaline, dopamine)
* Altered level of consciousness (Glasgow Coma Scale score < 13), repeated seizures, or status epilepticus
* Medical decision to limit treatment: no intubation, no admission to intensive care
* Refusal to participate in the study or participation in another interventional study on respiratory distress or acute respiratory failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with intubation criteria within 7 days | 7 days after randomization
  The proportion of patients requiring endotracheal intubation within 7 days after randomization. Intubation will be defined as the insertion of an endotracheal tube for invasive invasive mechanical ventilation

SECONDARY OUTCOMES:
All cause mortality at 28 days | 28 days after randomization
  Proportion of patients who have died from any cause within 28 days after randomization. Mortality will be assessed using medical records and/or direct patient follow-up
Organ failure-free days at 7 days | 7 days after randomization
  Organ failure will be defined using SOFA score or Modified SOFA score. The score ranges from 0 to 24.
CPAP tolerance Assessment | 7 days after intiation CPAP
  Patient discomfort will be assessed using a visual analog scale ranging from 0 (no discomfort) to 10 (maximum imaginable discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Armand Mekontso-dessap, professor, Study Chair — Assistance Publique - Hôpitaux de Paris; Ismael Guibla, doctor, Principal Investigator — University Hospital Souro Sanou, Burkina Faso; Ibrahim Alain Traore, professor, Study Director — University Hospital Souro Sanou, Burkina Faso
Locations (4):
- Burkina Faso (4):
  - Centre Hospitalier Universitaire Souro Sanou, Bobo-Dioulasso, Houet
  - CHU Yalgado Ouedraogo, Ouagadougou, Kadiogo
  - CHU Tengandogo, Ouagadougou, Kadiogo
  - CHU Bogodogo, Ouagadougou, Kadiogo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Markou NK, Myrianthefs PM, Baltopoulos GJ. Respiratory failure: an overview. Crit Care Nurs Q. 2004 Oct-Dec;27(4):353-79. doi: 10.1097/00002727-200410000-00006. PMID 15537123
- [Result] Stefan MS, Shieh MS, Pekow PS, Rothberg MB, Steingrub JS, Lagu T, Lindenauer PK. Epidemiology and outcomes of acute respiratory failure in the United States, 2001 to 2009: a national survey. J Hosp Med. 2013 Feb;8(2):76-82. doi: 10.1002/jhm.2004. Epub 2013 Jan 18. PMID 23335231
- [Result] SRLF Trial Group. Hypoxemia in the ICU: prevalence, treatment, and outcome. Ann Intensive Care. 2018 Aug 13;8(1):82. doi: 10.1186/s13613-018-0424-4. PMID 30105416
- [Result] Perkins GD, Ji C, Connolly BA, Couper K, Lall R, Baillie JK, Bradley JM, Dark P, Dave C, De Soyza A, Dennis AV, Devrell A, Fairbairn S, Ghani H, Gorman EA, Green CA, Hart N, Hee SW, Kimbley Z, Madathil S, McGowan N, Messer B, Naisbitt J, Norman C, Parekh D, Parkin EM, Patel J, Regan SE, Ross C, Rostron AJ, Saim M, Simonds AK, Skilton E, Stallard N, Steiner M, Vancheeswaran R, Yeung J, McAuley DF; RECOVERY-RS Collaborators. Effect of Noninvasive Respiratory Strategies on Intubation or Mortality Among Patients With Acute Hypoxemic Respiratory Failure and COVID-19: The RECOVERY-RS Randomized Clinical Trial. JAMA. 2022 Feb 8;327(6):546-558. doi: 10.1001/jama.2022.0028. PMID 35072713
- [Result] Templier F, Dolveck F, Baer M, Chauvin M, Fletcher D. [Laboratory testing measurement of FIO2 delivered by Boussignac CPAP system with an input of 100% oxygen]. Ann Fr Anesth Reanim. 2003 Feb;22(2):103-7. doi: 10.1016/s0750-7658(02)00859-6. French. PMID 12706763